CLINICAL TRIAL: NCT06095336
Title: Comparison of the Effectiveness of Telerehabilitation and Conventional Physiotherapy Program in Chronic Neck and Back Pain Seen in Caregivers of Individuals With Special Needs
Brief Title: Telerehabilitation and Conventional Physiotherapy Program for Caregivers of Individuals With Special Needs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burak Buğday, lecturer, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/85
Record Dates: First submitted 2023-09-20; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Telerehabilitation; Neck Pain
Keywords: individual with special needs; back pain
MeSH Terms: conditions — Neck Pain; Back Pain | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: In the study, which was planned as a randomized controlled study, participants were randomly divided into 3 groups.
Who Masked: Participant
Masking Description: Participants in the study did not know the group they belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telereahabilitation arm (Experimental): The group receiving telerehabilitation will be given a video CD containing the exercise program that will be changed every 3 weeks, and in the first week of each change program, daily sessions will be held collectively via video conferencing under the supervision of a physiotherapist. In the first 3 weeks of the 12-week exercise program, neck joint movements, neck stretching exercises and posture exercises will be given. Between weeks 4-6, in addition to the exercises in the first 3 weeks, cervical and scapular stabilization exercises will be given in the following weeks. In the following weeks, between weeks 7-9, 4-way strengthening exercises will be included in the program in addition to the exercises performed in the previous weeks. Cervical and scapular stabilization exercises and strengthening exercises will be performed in the following weeks between weeks 10-12, Exercises will be done 10 repetitions 3 times a day.
  Interventions: Other: telerehabilitation
- conventional physiotherapy arm (Experimental): Superficial heat (infrared), "Transcutaneous Electrical Nerve Stimulation" (TENS), therapeutic ultrasound and Hotpack application will be applied to the traditional treatment group. The patients receive 20 sessions in total, 5 days a week and 1 session daily for 4 weeks; You will receive superficial heat (infrared), TENS, therapeutic US and Hotpack treatment. . Superficial heat infrared will be applied to the tissue for 20 minutes. Conventional TENS will be applied. Therapeutic US will be applied to the cervical and thoracic region with an ultrasound device for 5 minutes at 3mHz, 1W/cm² treatment dosage, in continuous mode. Hotpack application will be done for 20 minutes. At the end of the 20 sessions, a brochure containing video-supported exercises will be given to the patients in the first group and they will be asked to do it for 12 weeks without follow-up.
  Interventions: Other: telerehabilitation
- control arm (No Intervention): The third group, the control group, will not receive any intervention and will be asked to continue their daily lives.

INTERVENTIONS:
Other: telerehabilitation — The individuals included in the research will be divided into three groups. Group 1 (experiment): This is the exercise group followed by the telerehabilitation method. Group 2 (experiment): This is the group where traditional physical therapy methods will be applied. The 3rd group will be taken as the control group, there will be no intervention and they will be asked to continue their daily lives.
  Other Names: conventional physiotherapy; control
  Arms: Telereahabilitation arm; conventional physiotherapy arm

SUMMARY:
The study was planned to investigate the effectiveness of home therapy method due to the difficulties experienced by caregivers of individuals with special needs in accessing physiotherapy and rehabilitation services for chronic neck and back pain.

DETAILED DESCRIPTION:
Caring for a disabled child is a very difficult and long process for parents. In this process, mothers and fathers exert a lot of effort while caring for the child, carrying the child and playing an active role in its rehabilitation. For these reasons, it is reported that the physical health of mothers and fathers is negatively affected and they often experience waist and back pain. Telerehabilitation allows patients who cannot access rehabilitation due to geographical, economic or physical disabilities to benefit from rehabilitation services. The distance problem is especially valid in cases where people live far from the rehabilitation center, there are no rehabilitation professionals specialized in the relevant disease in the place of residence, when transfers are difficult due to mobility problems, and in cases where it is not possible or risky to go to the rehabilitation center due to epidemics, as is the case today. Telerehabilitation has the potential to overcome all these problems. The study was planned to investigate the effectiveness of home therapy method due to the difficulties experienced by caregivers of individuals with special needs in accessing physiotherapy and rehabilitation services for chronic neck and back pain.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-60 years old,
* Being a special needs child caregiver,
* Mechanical neck and back pain lasting 3 months or longer

Exclusion Criteria:

* Those who are caregivers of hearing and visually impaired children,
* Having previously undergone surgery in the cervical region,
* Patients with a history of inflammatory or infective arthritis in the cervical spine,
* Congenital spinal cord anomaly,
* history of malignancy,
* Having neuropathic pain
* Radiculopathy, myelopathy or other neurological disorders
* Those with chronic lung disease
* Vestibular disorders,
* Those with a history of continuous drug use,
* Individuals who have been involved in an exercise or physiotherapy program in the last 3 months,
* He will not be able to read the scales and the evaluation parameters will be excluded from the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-28 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Demographic information form | before treatment
  The survey form prepared by the researcher in line with the literature includes information about the patients' name, surname, CV, family history, age, height, weight, occupation, dominant side, smoking and alcohol use, and additional symptoms.
Qualitative Questions Form | before treatment, after treatment, after 6 months
  A form containing questions asking about the number of individuals with special needs that they care for, the time they spend with the individual with special needs on a daily basis, the presence of another child other than the individual with special needs that they care for, whether there is help at home, the GMFCS Score of the individuals being cared for, and whether physical, mental or both effects are at the same time. will be prepared and implemented.
Pain Assessment | before treatment, after treatment, after 6 months
  Visual Analog Scale (VAS) was used to determine the severity of pain in the cases. The beginning will be marked as 0 (no pain) and the end (unbearable pain) on a 10 centimeter (cm) horizontal line, and the subjects will be asked to make a mark on this horizontal line according to the degree of pain they feel. The marked point on the line will then be measured with the help of a ruler and recorded as the VAS value in cm.
Fatigue Assessment: | before treatment, after treatment, after 6 months
  The FACIT Scale is a measurement tool consisting of 13 statements that subjectively evaluates fatigue in the last week. The scale has a five-point Likert scale: "0 = not at all, 1 = very little, 2 = a little, 3 = quite a bit and 4 = very much." 11 items (1-6, 9-13) of the scale contain reverse expressions. Items 7 and 8 of the scale are calculated as straight. The scores that can be obtained from the scale vary between 0-52. A high total score of the scale indicates that the severity of fatigue is low. If the score obtained from the scale is 30 or less, it is reported that perceived fatigue is clinically severe.
Short Form-36 (Short Form-36, SF-36): | before treatment, after treatment, after 6 months
  It is a valid and frequently used measure to evaluate quality of life. It includes 36 questions in eight subscales: physical function, physical role limitation, emotional role limitation, body pain, social function, mental health, vitality, and general health.

SECONDARY OUTCOMES:
Bournemouth Neck Pain Survey: | before treatment, after treatment, after 6 months
  It will be used to evaluate individuals with neck pain in terms of pain severity, participation in family and social life, depression, anxiety, kinesiophobia and pain coping skills. Individuals will be asked to give points between 0 and 10 for a total of 7 questions.
Caregiving Burden Scale: | before treatment, after treatment, after 6 months
  The Caregiving Burden Scale (CAÖ) is a 14-item scale. BYÖ's item scores are between 0-5. 0 means "Never", 1 means "Rarely", 2 means "Sometimes", 3 means "Often", and 4 means "Almost always". The evaluation of the ACO, in which all items are expressed plainly, is made on the basis of the total score.

CONTACTS AND LOCATIONS:
Overall Officials: burak buğday, Principal Investigator — Inonu University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terzi R, Tan G. Musculoskeletal system pain and related factors in mothers of children with cerebral palsy. Agri. 2016 Jan;28(1):18-24. doi: 10.5505/agri.2015.74436. PMID 27225608
- [Background] Hailey D, Roine R, Ohinmaa A, Dennett L. Evidence of benefit from telerehabilitation in routine care: a systematic review. J Telemed Telecare. 2011;17(6):281-7. doi: 10.1258/jtt.2011.101208. Epub 2011 Aug 15. PMID 21844172
- See also: pubmed — https://pubmed.ncbi.nlm.nih.gov/21844172/